CLINICAL TRIAL: NCT03792620
Title: A Conceptual Study of Daratumumab Intensified Treatment to Eligible Multiple Myeloma New Patients- Cyclophosphamide, Thalidomide, Dexamethasone and Daratumumab Induction, Follow by Daratumumab Consolidation and Maintenance
Brief Title: Daratumumab Intensified Treatment to Eligible MM New Patients CTD-Dara Induction, Follow by Dara Consolidation
Acronym: MAXDARA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Grupo de Estudos Multicentricos em Onco-Hematologia (Network)
Responsible Party: Principal Investigator, Edvan de Queiroz Crusoe, Gammopathy outpatient cordinator, Grupo de Estudos Multicentricos em Onco-Hematologia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1219-9010; CAAE (Other: 96591818.0.0000.0048)
Record Dates: First submitted 2018-11-19; First posted 2019-01-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Multiple Myeloma Stage I
Keywords: multiple myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Cyclo Thal Dex Daratumumab (Experimental): Eligible patients will be enrolled and treated according to the following elicited schema: Cyclo Thal Dex- Daratumumab (cyclophosphamide 500mg D1-8-15 + thalidomide 100-200mg D1-28 + dexamethasone 40mg/week (28 days cycle)- 4 cycles. ) + Daratumumab 16mg/Kg every week on cycles 1 and 2 and every other week at cycles 3 and 4- (total of 12 doses). Then Daratumumab 16mg/Kg after D+30, every other week as pre consolidation until starts full consolidation D+90-120 every other week (total of 4 doses) + thal100mg D1-28 during sixteen weeks as full consolidation. Follow by Daratumumab 16mg/Kg once a month as maintenance until progression or limiting adverse event (total of 28 planning doses).
  Total scheme Daratumumab doses= 50 doses = PROTOCOL MAXDARA.
  Interventions: Combination Product: Cyclo Thal Dex Daratumumab

INTERVENTIONS:
Combination Product: Cyclo Thal Dex Daratumumab — Cyclo Thal Dex Daratumumab
  Other Names: CTD-Dara,

SUMMARY:
The best induction protocol to eligible multiple myeloma patients was not established. Combination of three drugs demonstrated better outcomes than two drugs combo. Nevertheless, until now four drugs combo did not prove gain against three drugs One of the three drugs protocol studied as induction was CTD scheme (cyclophosphamide+ thalidomide+dexamethasone). Daratumumab has a novel mechanism of action that results in enhanced activity in combination with existing standards of care, including first-generation novel agents, such as thalidomide, as well as other therapeutics. Considerable responses have been observed in a cohort of heavily pretreated patients with relapsed/refractory MM. The use of a treatment combination with monoclonal antibody associated with immunomodulator (in a four drug combo) can lead to a improvement in response rates and in survival, reflects on a better free time interval. This trial will represent a new option of treatment with a combination of anti CD38 monoclonal antibody (DARATUMUMAB) as induction regimen with CTD protocol (four drug combination). And It use as consolidation and maintenance to give better immunomodulatory response and extended survival and disease control.

DETAILED DESCRIPTION:
Multiple Myeloma (MM) is a molecularly heterogeneous disease with a high degree of genomic instability. Despite improvements in event-free survival and overall survival with the use of autologous stem cell transplantation and novel agents, MM remains an incurable disease (1,2). The best induction protocol to eligible patients was not established. Combination of three drugs demonstrated better outcomes than two drugs combo. Nevertheless, until now four drugs combo did not prove gain against three drugs One of the three drugs protocol studied as induction was CTD scheme (cyclophosphamide+ thalidomide+dexamethasone) (3). This is an induction protocol commonly used in Brazil , with largely access in the brazilian public health system. Several new molecules have been developed in an attempt to improve treatment. One of these new treatment is an anti CD38 (Daratumumab). This potential target is present on plasma cells. The CD38 is a transmembrane glycoprotein recognized by combining several functions including adhesion, receptor and enzymatic function. (4-6) The expression of CD38 is finely regulated during ontogenesis of B cells and is expressed by progenitors and early stages hematopoietic cells with loss during maturation and only re- expressed during cellular activation .(4) With the information derived from tissue distribution and from pioneer experience in vitro indicates that very early precursors of the hematopoietic stem cells do not express CD38.(7) Despite the description of CD38 on progenitor cells, there was no myelosuppressive effect observed in studies to date. Apart from immune cells, the molecule CD38 has also been found in the brain, pancreatic acinar cells, smooth muscle and osteoclasts although expression in these tissues is in the cytosol or nucleus rather than the cell membrane. (8). Daratumumab has shown a strong signal in preclinical modeling with broad-spectrum killing activity through complement-mediated cytotoxicity (CDC), antibody-dependent cell-mediated cytotoxicity (ADCC), and ADC phagocytosis . (9) Daratumumab was first evaluated clinically in a phase I trial involving patients with relapsed/refractory multiple myeloma (10). In combination with others agents (lenalidomide + dexamethasone) preliminary analysis involving 20 patients, the rate of partial response or better was 75% with 3 patients achieving complete response and 6 patients a very good partial response (VGPR). The most common adverse reactions were infusion- related events (IREs) such as fever, cough, nausea, dizziness, and bronchospasm. A total of 9% occurred during predosing and 26% during the first full infusion with a gradual decrease with subsequent infusions. The onset of IREs was within 3-4 hours of infusion. Prophylactic steroids were administered to reduce the incidence of IREs (up to a maximum dose equivalent of 27 mg of dexamethasone per week). There were six serious adverse events (SAEs) related to daratumumab. Treatment-related adverse events included anemia, thrombocytopenia, and infusion reactions. All patients recovered from their SAEs with treatment and the maximum tolerated dose has not yet been reached. There was a dose-dependent decrease in peripheral-blood NK cells that was noted, with full recovery after treatment (11). Daratumumab has a novel mechanism of action that results in enhanced activity in combination with existing standards of care, including first-generation novel agents, such as thalidomide, as well as other therapeutics. Considerable responses have been observed in a cohort of heavily pretreated patients with relapsed/refractory MM. (12) However, in order to harness the full potential of the antimyeloma effect of daratumumab, the identification of synergistic drug combinations that target various mechanisms to overcome drug resistance will be vital. The potential role of cytotoxicity induced by the anti-CD38 antibody and the activation of effector cells with the immunomodulatory drugs could make this a very attractive antimyeloma combination therapy. Thalidomide, an oral immunomodulatory drug (IMID), has revolutionized clinical management of patients with MM with responses rates of 30% at relapse (alone) and higher rates at first line and at relapse when in combinations (50-65%) . The mechanism of action of thalidomide in myeloma cells remains under investigation. Thalidomide was found to potently inhibit the proliferation of endothelial cells and angiogenesis.

Thalidomide has direct cytotoxic effects on myeloma cells lines. In addition to its direct effect, IMIDs appear to modulate the bone marrow microenvironment. They can inhibit the up regulation of IL-6, necrose factor-α production and Vascular Endothelial Growth Factor (VEGF). It has a direct effect on the T-lymphocytes stimulating cytotoxic T cell proliferation, and induction of secretion of interferon γ and IL-2. The authors mentioned that as thalidomide does not show haematological toxicity, it may be used in advance disease when the platelet count is low . Thalidomide and the iMIDs have been used in combination with other chemotherapeutic agents with known and investigational activity in myeloma in several clinical trials. In vitro studies have suggested synergy between these agents and dexamethasone. The use of a treatment combination with monoclonal antibody associated with immunomodulator (in a four drug combo) can lead to a improvement in response rates and in survival, reflects on a better free time interval. Another interesting point is the use of Daratumumab intensified during consolidation and maintenance.

This trial will represent a new option of treatment with a combination of anti CD38 monoclonal antibody (Daratumumab) as induction regimen with CTD protocol (four drug combination). And It use as consolidation and maintenance to give better immunomodulatory response and extended survival and disease control.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have an Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2
* Participants who are newly diagnosed considered for high-dose chemotherapy due to: being age <=65 years; without presence of important comorbidity condition(s) likely to have a negative impact on tolerability of high dose chemotherapy with stem cell transplantation. Committee review and approval of participants is required before inclusion
* Women of childbearing potential must commit to either abstain continuously from sexual intercourse or to use 2 methods of reliable birth control simultaneously as deemed appropriate by the Investigator. Contraception must begin 4 weeks prior to dosing and must continue for 4 months after the last dose of DARATUMUMAB
* Man, who is sexually active with a woman of child-bearing potential potential must agree to use a latex or synthetic condom, even if he had a successful vasectomy, must agree to use an adequate contraception method as deemed appropriate by the Investigator, and must also agree to not donate sperm during the study and for four weeks after last dose of thalidomide and DARATUMUMB
* Participants with known or suspected COPD or asthma must have a FEV1 test during Screening

Exclusion Criteria:

* Participant has a diagnosis of primary amyloidosis, monoclonal gammopathy of undetermined significance (presence of serum M-protein <3 g/dL; absence of lytic bone lesions, anemia, hypercalcemia, and renal insufficiency related to the M-protein), or smoldering multiple myeloma (asymptomatic multiple myeloma with absence of related organ or tissue impairment end organ damage, and absence of biomarkers activity)
* Participant has a diagnosis of Waldenström's disease, or other conditions in which IgM M protein is present in the absence of a clonal plasma cell infiltration with lytic bone lesions
* Participant has a history of malignancy (other than multiple myeloma) within 5 years before the date of randomization (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy that in the opinion of the Investigator, with concurrence with the medical monitor, is considered cured with minimal risk of recurrence within 5 years)
* Participant has prior or current systemic therapy or SCT for multiple myeloma, with the exception of an emergency use of a short course (equivalent of dexamethasone 40 mg/day for a maximum 4 days) of corticosteroids 30 days before treatment
* Participant has had radiation therapy within 14 days of randomization
* Participant has known chronic obstructive pulmonary disease (COPD) (defined as a forced expiratory volume in 1 second [FEV1] <50% of predicted normal), persistent asthma, or a history of asthma within the last 2 years (controlled intermittent asthma or controlled mild persistent asthma is allowed)
* Participants with heart block defined by electrocardiogram or not treated arrhythmia
* Participant is known to be seropositive for history of human immunodeficiency virus (HIV) or known to have active hepatitis B or hepatitis C or Chagas disease positivity with cardiac involvement

Key exclusion criteria:

* Patient has malignancy , 3 years of first dose of study treatment (except basal or squamous cell carcinoma or in situ cancer of the cervix)
* Patients has not recovered from all therapy-related toxicities , grade 2 CTCAE; patients has undergone major surgery < 2 weeks prior to starting drug
* All patients must agree to follow the regional requirements for Thalidomide counseling, pregnancy testing and birth control. For women of childbearing potential (WOCBP) this includes pregnancy testing prior to prescribing thalidomide and to either commit to continued abstinence from heterosexual intercourse or begin acceptable methods of birth control for 28 days prior to prescribing thalidomide, during therapy and for 28 days after the last dose of thalidomide. WOCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a WOCBP even if they have had a successful vasectomy and must agree not to donate semen during study drug therapy and for a period of time after therapy. All patients must abstain from donating blood, agree not to share thalidomide with others and be counseled about the risks of thalidomide

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-11-20 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of response rate better than very good partial response after ASCT | 8 months after starting treatment
  Number of patients that obtained better than VGPR after ASCT based on the IMWG description

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE v 4.0 | 24 months
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0
Incidence of Overall response rate | 24 months
  Evaluate response rate as defined by the International Myeloma Working Group) IMWG- Minimal residual Disease (MRD), stringent complete Response (sCR), complete response (CR), very good partial response (VGPR), partial response (PR), and minimal response (MR) in patients treated with this protocol.
Duration of response after Dara-CTD treatment | 24 months
  Evaluate duration of response in patients treated with Daratumumab Cyclophosphamide thalidomide and dexamethasone treatment
Time of response after Dara-CTD treatment | 24 months
  Evaluate the specific moment of time of partial response observed after Daratumumab Cyclophosphamide thalidomide and dexamethasone treatment
Incidence of Minimal residual disease evaluate by PET CT image | 24 months
  Number of bone and extra bone marrow disease observed by PET CT image at diagnosis and after consolidation therapy by International Myeloma Working Group recommendations
Time to bone marrow engraftment | 24 months
  Measurement of neutrophil number in peripheral blood sample to evaluate the time of bone marrow engraftment
Number of progenitor cell collected after condition treatment | 24 months
  Flow cytometry of progenitor cell number collected
Time to Disease Progression (TTP). | 24 months
  Time to Disease Progression (TTP). The TTP is defined as time from date of randomization to date of first documented evidence of PD, as defined by IMWG criteria
Progression-Free Survival (PFS) and PFS on Next Line of Therapy (PFS2). | 24 months
  Progression-Free Survival (PFS) and PFS on Next Line of Therapy (PFS2).The PFS2 is defined as time from randomization to progression on next line of treatment or death, whichever occur first. Disease progression will be based on IMWG guide
Percentage of Participants With Negative Minimal Residual Disease (MRD). | 24 months
  The MRD assessment will be done by flow cytometry in bone marrow aspirate and in stem cell collected pack of participants four pre specified times- after induction, after ASCT, after consolidation and 1 year of maintenance
Peripheral blood lymphocytes number | 24 months
  Peripheral blood lymphocytes analysis will be done by Flow cytometry in spite of look at T and B population. The analysis will be performing at the same time as MRD
Time To Next treatment. | 24 months
  Time To Next treatment. Time to next treatment is defined as the time from randomization to the start of next-line treatment.
Duration of Response (DR). | 24 months
  Duration of Response (DR). The DR is time from date of initial documentation of response (PR or better) to date of first documented PD, as defined by IMWG criteria
Overall Survival (OS). | 24 months
  Overall Survival (OS). The OS is the time from date of randomization to date of participant's death or follow- up lost

CONTACTS AND LOCATIONS:
Overall Officials: Juliana Santos, Principal Investigator — CEHON
Locations (1):
- CEHON - Centro de Hematologia e Oncologia da Bahia, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Palumbo A, Anderson K. Multiple myeloma. N Engl J Med. 2011 Mar 17;364(11):1046-60. doi: 10.1056/NEJMra1011442. No abstract available. PMID 21410373
- [Result] Rajkumar SV, Dimopoulos MA, Palumbo A, Blade J, Merlini G, Mateos MV, Kumar S, Hillengass J, Kastritis E, Richardson P, Landgren O, Paiva B, Dispenzieri A, Weiss B, LeLeu X, Zweegman S, Lonial S, Rosinol L, Zamagni E, Jagannath S, Sezer O, Kristinsson SY, Caers J, Usmani SZ, Lahuerta JJ, Johnsen HE, Beksac M, Cavo M, Goldschmidt H, Terpos E, Kyle RA, Anderson KC, Durie BG, Miguel JF. International Myeloma Working Group updated criteria for the diagnosis of multiple myeloma. Lancet Oncol. 2014 Nov;15(12):e538-48. doi: 10.1016/S1470-2045(14)70442-5. Epub 2014 Oct 26. PMID 25439696
- [Result] Morgan GJ, Davies FE, Gregory WM, Bell SE, Szubert AJ, Navarro Coy N, Cook G, Feyler S, Johnson PR, Rudin C, Drayson MT, Owen RG, Ross FM, Russell NH, Jackson GH, Child JA; National Cancer Research Institute Haematological Oncology Clinical Studies Group. Cyclophosphamide, thalidomide, and dexamethasone as induction therapy for newly diagnosed multiple myeloma patients destined for autologous stem-cell transplantation: MRC Myeloma IX randomized trial results. Haematologica. 2012 Mar;97(3):442-50. doi: 10.3324/haematol.2011.043372. Epub 2011 Nov 4. PMID 22058209
- [Result] Sondergeld P, van de Donk NW, Richardson PG, Plesner T. Monoclonal antibodies in myeloma. Clin Adv Hematol Oncol. 2015 Sep;13(9):599-609. PMID 26452191
- [Result] Deaglio S, Mehta K, Malavasi F. Human CD38: a (r)evolutionary story of enzymes and receptors. Leuk Res. 2001 Jan;25(1):1-12. doi: 10.1016/s0145-2126(00)00093-x. PMID 11137554
- [Result] Reinherz EL, Kung PC, Goldstein G, Levey RH, Schlossman SF. Discrete stages of human intrathymic differentiation: analysis of normal thymocytes and leukemic lymphoblasts of T-cell lineage. Proc Natl Acad Sci U S A. 1980 Mar;77(3):1588-92. doi: 10.1073/pnas.77.3.1588. PMID 6966400
- [Result] Verfaillie CM, Miller JS. CD34+/CD33- cells reselected from macrophage inflammatory protein 1 alpha+interleukin-3--supplemented "stroma-noncontact" cultures are highly enriched for long-term bone marrow culture initiating cells. Blood. 1994 Sep 1;84(5):1442-9. PMID 7520771
- [Result] Phipps C, Chen Y, Gopalakrishnan S, Tan D. Daratumumab and its potential in the treatment of multiple myeloma: overview of the preclinical and clinical development. Ther Adv Hematol. 2015 Jun;6(3):120-7. doi: 10.1177/2040620715572295. PMID 26137203
- [Result] Laubach JP, Richardson PG. CD38-Targeted Immunochemotherapy in Refractory Multiple Myeloma: A New Horizon. Clin Cancer Res. 2015 Jun 15;21(12):2660-2. doi: 10.1158/1078-0432.CCR-14-3190. Epub 2015 Apr 15. PMID 25878332
- [Result] van de Donk NW, Lokhorst HM. New developments in the management and treatment of newly diagnosed and relapsed/refractory multiple myeloma patients. Expert Opin Pharmacother. 2013 Aug;14(12):1569-73. doi: 10.1517/14656566.2013.805746. Epub 2013 May 31. PMID 23721099
- [Result] Lonial S, Weiss BM, Usmani SZ, Singhal S, Chari A, Bahlis NJ, Belch A, Krishnan A, Vescio RA, Mateos MV, Mazumder A, Orlowski RZ, Sutherland HJ, Blade J, Scott EC, Oriol A, Berdeja J, Gharibo M, Stevens DA, LeBlanc R, Sebag M, Callander N, Jakubowiak A, White D, de la Rubia J, Richardson PG, Lisby S, Feng H, Uhlar CM, Khan I, Ahmadi T, Voorhees PM. Daratumumab monotherapy in patients with treatment-refractory multiple myeloma (SIRIUS): an open-label, randomised, phase 2 trial. Lancet. 2016 Apr 9;387(10027):1551-1560. doi: 10.1016/S0140-6736(15)01120-4. Epub 2016 Jan 7. PMID 26778538
- [Derived] de Queiroz Crusoe E, Leal Ribeiro Dos Santos JS, de Andrade Santos J, de Melo Santos HH, de Souza Santos A, Lucas LF, Requiao de Pinna CA, Caldas Freire PN, Araujo de Jesus A, de Moura Almeida A, Dutra DD, Chaves MF, Nicanor JS, Salvino MA, Bomfim Arruda MDG, Hungria V; GBRAM. Phase 2 trial of daratumumab, cyclophosphamide, thalidomide, and dexamethasone in newly diagnosed multiple myeloma. Blood Neoplasia. 2025 Mar 3;2(3):100081. doi: 10.1016/j.bneo.2025.100081. eCollection 2025 Aug. PMID 40575076